CLINICAL TRIAL: NCT02596386
Title: Examination of Potassium Levels in Saliva in ESRD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: k001.HMO-CTIL
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- potassium level in saliva: Each willing participant will undergo Sialometry
  Interventions: Procedure: sialometry
- blood test: blood will be drawn from the dialysis connections for Biochemistry for potassium level evaluation
  Interventions: Procedure: blood test

INTERVENTIONS:
Procedure: sialometry — potassium evaluation
  Groups: potassium level in saliva
Procedure: blood test — potassium evaluation
  Groups: blood test

SUMMARY:
Dialysis patients typically undergo 3 treatments a week every other day with an almost 3 day gap during the weekend. After this gap and before the first dialysis of the week the serum Potassium level is expected to be maximal.

Participants will be recruited from the dialysis clinic at Hadassah Ein Kerem Hospital. The research team would personally meet the patients who answer inclusion criteria f and ask whether they wish to participate.

Each willing participant will undergo Sialometry and blood will be drawn from the dialysis connections for CBC and Biochemistry to establish a baseline.

The study measurements namely Sialometry and collection of Saliva as well as blood test will be taken before the initiation of the dialysis.

Blood testing will be done via the laboratories of the Hadassah hospital. Saliva analysis will be done in the research lab of Prof. Doron Aframian.

ELIGIBILITY:
Inclusion Criteria:

* Present a predialysis serum potassium level over 5 mmol/L.

Exclusion Criteria:

* Pregnancy

Patients diagnosed with a pathology of the salivary glands such as Sjogren's syndrome, Sialosis, Sialadenitis.

Patients who have received previous radiation therapy to the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients on Hemodialysis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
potassium level in saliva | 7 days
Standard Biochemistry of blood | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Doron J Aframian, MD,PhD, Principal Investigator — Hadassah Medical Organization

REFERENCES:
- [Background] Seethalakshmi C, Koteeswaran D, Chiranjeevi V. Correlation of Serum and Salivary Biochemical Parameters in end Stage Renal Disease Patients Undergoing Hemodialysis in Pre and Post-Dialysis State. J Clin Diagn Res. 2014 Dec;8(12):CC12-4. doi: 10.7860/JCDR/2014/10404.5306. Epub 2014 Dec 5. PMID 25653941
- [Background] Davidovich E, Davidovits M, Peretz B, Shapira J, Aframian DJ. Elevated salivary potassium in paediatric CKD patients, a novel excretion pathway. Nephrol Dial Transplant. 2011 May;26(5):1541-6. doi: 10.1093/ndt/gfq587. Epub 2010 Oct 4. PMID 20921301